CLINICAL TRIAL: NCT04776980
Title: Multimodality MRI for Quantification of Tumor-associated Macrophages and Prediction of Somatic Mutation Detectability in Cell-free DNA in Adult Patients With Glioblastoma
Brief Title: Multimodality MRI and Liquid Biopsy in GBM
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI decision to close study
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Ali Nabavizadeh, Assistant Professor of Radiology at the Hospital of the University of Pennsylvania, Abramson Cancer Center at Penn Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 843601
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Glioblastoma Multiforme; Brain Tumor, Adult: Glioblastoma; Brain Tumor, Recurrent; Brain Tumor, Primary
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ferumoxytol Infused MRI (Experimental): Ferumoxytol is an iron replacement product that is FDA approved to treat iron deficiency anemia in patients with chronic kidney disease (CKD). In this study, ferumoxytol is used to quantify tumor-associated macrophages. The infused dose would be 5mg/kg.
  Interventions: Diagnostic Test: Post Feraheme Infusion MRI

INTERVENTIONS:
Diagnostic Test: Post Feraheme Infusion MRI — All participants will receive a ferumoxtyol (Feraheme) infusion 20-28 hours prior to a head MRI. In addition, a blood draw for liquid biopsy targeted tissue sampling during surgery and special iron and macrophage staining on the tumor tissue.

SUMMARY:
Patients with a new diagnosis of high-grade glioma based on MRI, who are considered surgical candidates determined by neurosurgeons or patients with recurrent glioblastoma with the initial diagnosis of glioblastoma (histologic or molecular proof) and recommended for clinically surgical resection may be eligible for this study. Subjects may participate in this study if they are at least 18 years of age.

Ferumoxytol-enhanced MRI will be used to quantify tumor-associated macrophages. This is a non-therapeutic trial in that imaging will not be used to direct treatment decisions.

The blood draw is being completed to evaluate cell-free circulating tumor DNA (cfDNA) and cell-free tumor DNA (ctDNA).

DETAILED DESCRIPTION:
This is a pilot study in subjects with a new diagnosis of high-grade glioma based on classic MRI appearance who are considered surgical candidates and patients with histologically proven diagnosis of glioblastoma (GB) who have completed chemoradiation and now have new contrast-enhancing lesions or lesions showing increased enhancement ( 25% increase) who are recommended for a clinical surgical resection. Subjects may participate in this study if they are at least 18 years of age, most participants will be receiving care at the clinical practices of the University of Pennsylvania. Subjects who come to the University of Pennsylvania for diagnosis and/or treatment of GB and who meet the study inclusion criteria may be approached by study personnel for recruitment into this study. Subjects will be approached about study participation regardless of race or ethnic background. Investigators anticipate enrolling up to 30 participants. Subjects who consent but do not complete the study imaging will be considered not evaluable and will be replaced. Accrual will likely occur over approximately 2 years. After undergoing screening assessments and verifying eligibility for study participation subjects will undergo a research ferumoxytol-enhanced MRI of the brain and blood draws for liquid biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be ≥ 18 years of age
2. Patients with new diagnosis of high grade glioma based on MRI, who are considered surgical candidates determined by neurosurgeons or recurrent glioblastoma with the initial diagnosis of glioblastoma (histologic or molecular proof) and recommended for clinically surgical resection
3. Life expectancy of greater than 3 months in the opinion of an investigator or treating physician.
4. Karnofsky performance status ≥ 60

Exclusion Criteria:

1. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
2. Females who are pregnant or breast feeding at the time of screening will not be eligible for this study; pregnancy status will be confirmed verbally prior to participating in any study procedures.
3. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study
4. Contraindications to MRI or use of ferumoxytol or gadolinium contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06-22 (Estimated)

PRIMARY OUTCOMES:
Macrophage quantification status | 2 years
  Macrophage quantification status will be determined using histology methods based on biopsy sites and will be correlated with ferumoxytol-enhanced MRI.

SECONDARY OUTCOMES:
Cell free tumor DNA (ctDNA) | 2 years
  To determine the proportion of mutations identified by biopsy that are correctly identified in samples of plasma ctDNA for each subject, and to explore the potential of imaging measures to predict that proportion

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Ali Nabavizadeh, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No